CLINICAL TRIAL: NCT04755374
Title: Clinical Characteristics and Discharge Assessment of Patients in a Recent Founded Palliative Care Unit
Brief Title: Clinical Characteristics and Discharge Assessment of Patients From Palliative Care
Status: Completed | Type: Observational
Sponsor: Diskapi Yildirim Beyazit Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Gulten Utebey, Dr, Diskapi Yildirim Beyazit Education and Research Hospital
Other Study IDs: Palliative-Discharge
Record Dates: First submitted 2021-02-11; First posted 2021-02-16 (Actual); Last update posted 2021-07-14 (Actual); Status verified 2021-02

CONDITIONS: Critical Illness
Keywords: Critical illness; Palliative care; Length of stay
MeSH Terms: conditions — Critical Illness | interventions — Drainage

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: Discharged from palliative care unit in equal or less than 21 days
  Interventions: Other: Discharged ≤ 21 days
- Group 2: Prolonged discharged in longer than 21 days: Discharged from palliative care unit in longer than 21 days
  Interventions: Other: Prolonged discharge

INTERVENTIONS:
Other: Discharged ≤ 21 days — Discharged from palliative care unit in equal less than 21 days
  Groups: Group 1
Other: Prolonged discharge — Discharged from palliative care unit in longer than 21 days
  Groups: Group 2: Prolonged discharged in longer than 21 days

SUMMARY:
The number of people having chronic diseases and the demand for palliative care has increased. The factors that have an impact on length of stay and discharge of patient who were admitted to palliative care center will be investigated.

DETAILED DESCRIPTION:
Adult patients admitted to the Diskapi Yildirim Beyazit Teaching and Research Hospitals Palliative Care Unit between August 2018 and September 2020 and discharged to their home will be retrospectively evaluated.

Patient's age, gender, diagnosis, conditions/comorbidities, Karnofsky Performance Scale, discharge status (death, intensive care unit or at home), gastrostomy status, presence of tracheostomy and/or mechanical ventilation, nutritional status (total parenteral nutrition or enteral nutrition), pressure ulcers, the lowest and highest recorded hemoglobin concentration, white blood cell count and serum sodium concentration and the education level of the patient and the caregiver will be recorded. Patients will be grouped according to length of stay (LOS) as Group 1: discharged in equal or less than 21 days or Group 2: Prolonged discharged in longer than 21 days and analysed accordingly

ELIGIBILITY:
Inclusion Criteria:

• Adult patients admitted to the palliative care unit

Exclusion Criteria:

• Patients not consenting to participate the study

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with a critical ilness/conditions
Sampling Method: Non-Probability Sample
Enrollment: 103 (Actual)
Dates: Start 2021-02-20 (Actual); Primary Completion 2021-03-20 (Actual); Study Completion 2021-04-20 (Actual)

PRIMARY OUTCOMES:
Length of stay | 24 hours after discharge
  Length of stay will be determined after discharge

CONTACTS AND LOCATIONS:
Overall Officials: Gulten Utebey, Dr, Principal Investigator — Ministry of Health
Locations (1):
- Diskapi Yildirim Beyazit Teaching and Research Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gomes B, Higginson IJ. Where people die (1974--2030): past trends, future projections and implications for care. Palliat Med. 2008 Jan;22(1):33-41. doi: 10.1177/0269216307084606. PMID 18216075
- [Background] Lau F, Downing GM, Lesperance M, Shaw J, Kuziemsky C. Use of Palliative Performance Scale in end-of-life prognostication. J Palliat Med. 2006 Oct;9(5):1066-75. doi: 10.1089/jpm.2006.9.1066. PMID 17040144
- [Background] Kelly A, Conell-Price J, Covinsky K, Cenzer IS, Chang A, Boscardin WJ, Smith AK. Length of stay for older adults residing in nursing homes at the end of life. J Am Geriatr Soc. 2010 Sep;58(9):1701-6. doi: 10.1111/j.1532-5415.2010.03005.x. Epub 2010 Aug 24. PMID 20738438